CLINICAL TRIAL: NCT02485496
Title: SECURE - A poSt-market Registry in Patients With infrarEnal aortiC Aneurysm Undergoing endovasculaR Stenting With the New E-tegra Stent Graft System
Brief Title: E-tegra Stent Graft System in the Treatment of Infra-renal Abdominal Aortic Aneurysms
Acronym: SECURE
Status: Terminated | Type: Observational
Why Stopped: Due to product change.
Sponsor: JOTEC GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: SECURE
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Abdominal Aortic Aneurysm; AAA
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Endovascular abdominal repair
  Other Names: EVAR

SUMMARY:
The purpose of this study is to evaluate clinical and technical success as well as safety and feasibility of the E-tegra Stent Graft System used in endovascular treatment of infrarenal aortic aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* Patients must comply with the indications for use
* Patient must have an infrarenal aortic aneurysm with diameter >5cm or an infrarenal aortic aneurysm with 4 to 5cm that has increased in size by 0.5cm in the last 6 months
* Patient must be available for the appropriate follow-up times for the duration of the study
* Patient has signed the informed consent before intervention

Exclusion Criteria:

* Patients with one of the contraindications as indicated in the instructions for use
* Patients with infectious aneurysm
* Patients with inflammatory aneurysm
* Patients with pseudoaneurysm
* Patients with ruptured or traumatic aneurysm
* Patients with suprarenal, juxtarenal, or pararenal aneurysm
* Patients with aortic dissection
* Patients with a reversed conical neck that is defined as a >3mm distal increase over a 15mm length
* Patients who have a congenital degenerative Collagen disease or connective tissue disorder
* Patients with thrombocytopenia
* Patients with creatinine >2.4 mg/dl immediately before the Intervention
* Patients with hyperthyreosis
* Patients with malignancy needing chemotherapy or Radiation
* Patients who are enrolled in another clinical study
* Patients with life expectancy of less than 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with infrarenal aortic or aorto-iliac aneurysm who are eligible for treatment with an abdominal stent graft according to the instructions for use for the E-tegra stent graft system, and scheduled for implantation of the E-tegra stent graft system at their physician's discretion in accordance with the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-06; Primary Completion 2020-07 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Rate of aneurysm rupture and aneurysm related death | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sven Seifert, Dr., Principal Investigator — Klinikum Chemnitz
Locations (10):
- France (2):
  - CHU Nantes, Nantes
  - CHU Pontchaillou, Rennes
- Germany (2):
  - Klinikum Chemnitz, Chemnitz
  - Universitätsklinikum Leipzig, Leipzig
- Poland (3):
  - Szpital Uniwersytecki im. dr. Antoniego Jurasza, Bydgoszcz
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Lublin
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
- Spain (2):
  - Hospital Joan XXIII, Tarragona
  - Hospital Clinico Universitario Valladolid, Valladolid
- Inselspital - Universitätsspital, Bern, Switzerland